CLINICAL TRIAL: NCT00157859
Title: To Evaluate the Efficacy of Chloroquine and SP for Acute Uncomplicated P. Falciparum and the Efficacy of Chloroquine for Acute Uncomplicated P. Vivax in the Timika Region of Papua, Indonesia.
Brief Title: To Evaluate Current Efficacy of Antimalarials Used in Timika, Papua, Indonesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menzies School of Health Research (Other)
Collaborators: Wellcome Trust (Other); National Health and Medical Research Council, Australia (Other); National Institute of Health Research and Development, Ministry of Health Republic of Indonesia (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Timika_FP_VP; Wellcome Trust ME028458MES
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2005-09

CONDITIONS: Falciparum Malaria; Vivax Malaria
Keywords: Falciparum; Vivax; Papua; Chloroquine; Sulphadoxine-pyrimethamine
MeSH Terms: conditions — Malaria, Falciparum; Malaria, Vivax | interventions — Chloroquine; fanasil, pyrimethamine drug combination

INTERVENTIONS:
Drug: Chloroquine and sulphadoxine-pyrimethamine

SUMMARY:
Multidrug resistant strains of P.falciparum and P.vivax are becoming increasingly prevalent in the Asia Pacific rim. To determine the efficacy of locally recommended antimalarial protocols in Papua, Indonesia, consecutive patients presenting to a rural clinic were enrolled into a prospective efficacy study. Patients with uncomplicated falciparum malaria were treated with chloroquine plus sulfadoxine-pyrimethamine and those with vivax malaria with chloroquine monotherapy. Patients failing therapy received unsupervised oral quinine +/- doxycycline for 7 days. Follow-up was continued for 42 days for falciparum malaria and 28 days for vivax malaria.

The study hypothesis was that current recommended antimalarial protocols were no longer effective.

ELIGIBILITY:
Inclusion Criteria:

-Male and female patients at least one 1year of age and weighing more than 10kg.

* -Microscopic confirmation of P. falciparum and /or P.vivax infection (any parasitaemia).
* -Fever (axillary temperature >37.5oC) or history of fever in the last 48 hours.
* -Able to participate in the trial and comply with the clinical trial protocol
* -Written informed consent to participate in trial; verbal consent in presence of literate witness is required for illiterate patients, and written consent from parents/guardian for children below age of consent

Exclusion Criteria:

* Pregnancy or lactation

  * -Inability to tolerate oral treatment
  * -Signs/symptoms indicative of severe/complicated malaria or warning signs requiring parenteral treatment
  * -Known hypersensitivity or allergy to artemisinin derivatives
  * -Serious underlying disease (cardiac, renal or hepatic)
  * -Parasitaemia >4%

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150
Dates: Start 2004-04; Study Completion 2004-09

PRIMARY OUTCOMES:
• 42 day cure rate; corrected for reinfection by PCR genotyping.
• Overall Cure Rate at Day 42

SECONDARY OUTCOMES:
• Overall day 28 cure rate for P.falciparum. This will allow comparison with previous historical data at this time point.
• Parasite reduction. Parasite reduction will be calculated at Days 1, 2 and 3 after initiation of trial treatment as percentage of parasites/uL compared to parasite density before the first dose of treatment.
• Proportion of patients with a negative slide at Days 1, 2 and 3
• Gametocyte Carriage. Anti-gametocyte activity will be measured by the proportion of patients with a peripheral gametocytaemia between day 7 to day 28.
• Early Treatment Failure (ETF)
• Late Treatment Failure (LTF)

CONTACTS AND LOCATIONS:
Overall Officials: Emiliana Tjitre, PhD, Principal Investigator — National Institute of Health Research and Development, Ministry of Health Republic of Indonesia
Locations (1):
- SP9 & SP12 Public Health- Malaria control clinics, Timika, Special Region of Papua, Indonesia